CLINICAL TRIAL: NCT02716168
Title: Partnership-Project - Reinforcing Partnership Between Cancer Patient, General Practitioner and Oncologist During Chemotherapy - a Randomized Controlled Trial
Brief Title: Partnership-Project - Reinforcing Partnership Between Cancer Patient, General Practitioner and Oncologist During Chemotherapy
Acronym: PSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Research Center of Cancer Rehabilitation (Unknown); Research Unit of General Practice, Odense (Other); Vejle Hospital (Other); Region of Southern Denmark (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Theis Trabjerg, MD, PhD fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Partnership-Project
Record Dates: First submitted 2016-03-03; First posted 2016-03-23 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cancer
Keywords: Cancer; tele-health; Shared care; Continuity
MeSH Terms: conditions — Neoplasms | interventions — General Practitioners; Oncologists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Video consultation (Experimental): Video consultation between cancer patient, general practitioner and oncologist at the start of chemotherapy treatment
  Interventions: Other: Shared video consultation between patient, general practitioner and oncologist
- usual care (No Intervention): Usual care. The patients General Practitioner will receive standard discharge summary and ambulant notes from the oncologist specialist

INTERVENTIONS:
Other: Shared video consultation between patient, general practitioner and oncologist — At the start of the patients chemotherapy treatment a shared video consultation between the patient, general practitioner and oncologist will bee arranged. The video consultation should address distribution of roles, comorbidity, medicine, depression and anxiety symptoms, relatives and social resources.
  Arms: Video consultation

SUMMARY:
Background International guidelines underline the importance of strengthening the coordination and continuity of cancer care. The different roles of general practitioners and oncologists with regard to treatment, follow-up and rehabilitation during and after cancer treatment are often obscure to cancer patients. Parallel courses of healthcare are often taking place instead of coordinated care characterized by continuity and partnership between care providers. Patients may feel uncertain about the health professionals' skills and area of responsibility. Healthcare seeking and support during and after cancer treatment may, therefore, be inappropriate, leaving patients feeling insecure and lost between care providers.The study aims to design and evaluate a new way of communication and shared decision-making that brings the patient, the oncologist and general practitioner together in a shared video-consultation in the early phase of chemotherapeutic treatment. The effect of the intervention in addition to usual care will be tested in a randomized controlled trial at Vejle Hospital in the Region of Southern Denmark. Based on sample size calculation, investigators intent to include 300 patients at the Department of Oncology and their general practitioners. Results and process outcomes will be evaluated qualitatively and quantitatively, questionnaires to patients, general practitioners and oncologists, and data from registers.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred cancer patient scheduled for chemotherapy at the Department for Oncology, Vejle Hospital, Region of Southern Denmark
* Aged 18 years and over
* Able to speak and read Danish
* Mentally able to cooperate
* Listed with a general practitioner (98 % of the danish population)
* Written and verbal informed consent given

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Shared Care questionnaire | 7 month after inclusion
  Patient reported outcome measure. Cancer patients assessment of their cancer trajectory and their assessment of the cooperation between their General Practitioner and the oncologist specialist.

SECONDARY OUTCOMES:
Illness Intrusiveness Rating Scale (IIRS) | 4 and 7 month after inclusion
  Patient reported outcome measure. Patients assessment of the cancer disease influence on their daily living.
European Organisation for Research and Treatment of Cancer - Quality of Life questionnaire - Core 30 (EORTC QLQ C30) | 4 and 7 month after inclusion
  Patient reported outcome measure. Cancer patients assessment of their quality of life
European Organisation for Research and Treatment of Cancer - Quality of Life- information questionnaire (EORTC QLQ INFO25) | 4 and 7 month after inclusion
Generalised Anxiety Disorder Assessment (GAD-7) | 4 and 7 month after inclusion
  Patient reported outcome measure. Screening tool and severity measure for generalised anxiety disorder
Patient Health Questionnaire (PHQ-9) | 4 and 7 month after inclusion
  Patient reported outcome measure.The questionnaire monitor the severity of depression and response to treatment.
Oncologist assessment of a video consultation between the patient, General practitioner and oncologist. | Directly after the video consultation intervention
  It measures the oncologist perception of the benefits with the video consultation intervention. Only the intervention group
General practitioners assessment of a video consultation between the patient, General practitioner and oncologist. | Directly after the video consultation intervention
  It measures the General Practitioners perception of the benefits with the video consultation intervention. Only the intervention group.
Patients assessment of a video consultation between the patient, General practitioner and oncologist. | Directly after the video consultation intervention
  It measures the patients perception of the benefits with the video consultation intervention.Only the intervention group
General Practitioner cancer trajectory assessment | 4 month after the inclusion of the patient.
  The General Practitioners assessment of the cooperation between the primary and secondary care regarding af specific cancer patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Vejle Hospital, Region of Southern Denmark, Vejle, Denmark

REFERENCES:
- [Derived] Baygi F, Trabjerg TB, Jensen LH, Munch Storsveen M, Wehberg S, Sondergaard J, Gilsa Hansen D. Impact of Cross-Sectoral Video Consultation on Perceived Care Coordination and Information Satisfaction in Cancer Care: Randomized Controlled Trial. JMIR Form Res. 2025 Dec 31;9:e76910. doi: 10.2196/76910. PMID 41474977
- [Derived] Hansen DG, Trabjerg TB, Sisler JJ, Sondergaard J, Jensen LH. Cross-sectoral communication by bringing together patient with cancer, general practitioner and oncologist in a video-based consultation: a qualitative study of oncologists' and nurse specialists' perspectives. BMJ Open. 2021 May 5;11(5):e043038. doi: 10.1136/bmjopen-2020-043038. PMID 33952540
- [Derived] Trabjerg TB, Jensen LH, Sondergaard J, Sisler JJ, Hansen DG. Cross-sectoral video consultations in cancer care: perspectives of cancer patients, oncologists and general practitioners. Support Care Cancer. 2021 Jan;29(1):107-116. doi: 10.1007/s00520-020-05467-0. Epub 2020 Apr 21. PMID 32318872
- [Derived] Trabjerg TB, Jensen LH, Sondergaard J, Sisler JJ, Hansen DG. Improving continuity by bringing the cancer patient, general practitioner and oncologist together in a shared video-based consultation - protocol for a randomised controlled trial. BMC Fam Pract. 2019 Jun 25;20(1):86. doi: 10.1186/s12875-019-0978-8. PMID 31238886